CLINICAL TRIAL: NCT06789497
Title: Lovastatin Modulation of the Inhibition-excitation Balance in Temporal Lobe Onset Drug Resistant Epilepsy
Brief Title: The GABAergic Inhibitory System in Drug Resistant Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Miguel Castelo-Branco, Prof Dr, University of Coimbra
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CIBIT-EPILEPSY-1; FLAD Life Science 2020 (Other Grant/Funding Number: Luso-American Development Foundation)
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Drug Resistant Epilepsy; Temporal Lobe Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy, Temporal Lobe | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lovastatin (Experimental)
  Interventions: Drug: Lovastatin 60 MG
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovastatin 60 MG — Participants were given lovastatin 60 mg/day for three consecutive days.
  Arms: Lovastatin
Drug: Placebo — Participants were given placebo 60 mg/day for three consecutive days.
  Arms: Placebo

SUMMARY:
This study aims to investigate the effect of lovastatin on neurotransmission and neuroinflammation in patients with temporal lobe onset drug resistant epilepsy.

Structure: (1) Visit 1: 3 consecutive days of physiologically probing drug/placebo intake, (2) Visit 2: Outcome measures and additional evaluations in the day after the last drug/placebo intake, (3) Washout period of 4 weeks, (4) 3 consecutive days of drug/placebo intake, (5) Visit 3: Outcome measures and additional evaluations in the day after the last placebo/drug intake.

DETAILED DESCRIPTION:
This study investigates the potential therapeutic effects of lovastatin, a drug known for its anti-inflammatory and neuroprotective properties, in patients with temporal lobe drug-resistant epilepsy (DRE). Emerging evidence suggests that inflammation plays a significant role in epileptogenesis, and preclinical models of epilepsy have demonstrated the efficacy of statins in reducing seizure susceptibility.

This pilot, double-blinded, placebo-controlled crossover study included five participants with focal-onset DRE. The primary objectives were to evaluate the impact of lovastatin on cortical inhibition, oxidative stress, and seizure activity. Participants received 60 mg/day of lovastatin or placebo for a specified period, with treatment phases separated by a washout period.

Key assessments included magnetic resonance spectroscopy (MRS) to measure brain metabolites such as GABA, glutamate, and glutathione in the occipital cortex. Event-related potentials (ERP) were recorded during a facial recognition task to examine visual evoked potentials, while resting EEG was used to analyze interictal epileptiform discharges (IEDs).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pharmacoresistant epilepsy as defined by the International League Against Epilepsy,
* focal temporal lobe onset
* nonpregnant and nonlactating in women

Exclusion Criteria:

* history of cardiovascular or cerebrovascular disease,
* history of dyslipidemia, previous use of statins or a previously documented adverse reaction to statins,
* having any metal inside the head but outside the mouth,
* implanted devices such as cardiac pacemakers or cochlear implants,
* having a vagal nerve stimulation device and the presence of other comorbid neurologic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Neurochemical response changes to GABAergic stimulation | First day after placebo and first day after lovastatin intervention.
  Comparing changes in brain excitation-inhibition measures (i.e., glutamate and GABA) when the GABAergic system is activated by oral dose of the Lovastatin 60mg during 3 days versus the placebo condition.
Evaluation of neuroinflammation by measuring Glutathione as a marker of oxidative stress | First day after placebo and first day after lovastatin intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nuclear Sciences Applied to Health, Coimbra, Coimbra District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided